CLINICAL TRIAL: NCT01323088
Title: Physical Activity in Overweight Girls: Implications for Reversing Risk Factors for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R21DK083654-01A1 (NIH)
Record Dates: First submitted 2011-03-22; First posted 2011-03-25 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Abdominal Obesity; Physical Activity
Keywords: Childhood obesity; Visceral fat; Insulin resistance; Liver fat; Skeletal muscle lipid; Regular exercise
MeSH Terms: conditions — Obesity, Abdominal; Motor Activity; Pediatric Obesity; Insulin Resistance; Fatty Liver | interventions — Resistance Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Other): Standard care control (no-exercise)
  Interventions: Other: Control
- Aerobic Exercise (Active Comparator)
  Interventions: Other: Aerobic exercise
- Resistance Exercise (Active Comparator)
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Other: Control — Standard care control (no exercise)
  Arms: Control
Other: Resistance Exercise — Supervised resistance exercise using stack weight equipments.
  Arms: Resistance Exercise
Other: Aerobic exercise — Supervised aerobic exercise using treadmills, bikes, and ellipticals
  Arms: Aerobic Exercise

SUMMARY:
In this randomized controlled trial, we will examine the effect of a 3-month exercise training (aerobic exercise versus resistance exercise) without calorie restriction on total and regional adiposity, ectopic fat in the liver and skeletal muscle, and risk of type 2 diabetes in overweight girls.

ELIGIBILITY:
Inclusion Criteria:

* Healthy overweight (BMI >-95th) youth between 12 and 18 years of age
* Waist circumference >-75th percentile
* Sedentary (no structured exercise >2 times/week for past 6 months)
* Non-smokers, non-diabetic, no medical conditions
* Weight stable for past 3 months

Exclusion Criteria:

* Smokers
* Diabetes
* Psychiatric disorders
* Syndromic obesity
* Pregnancy
* Taking medications known to affect study outcomes

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Abdominal obesity, visceral fat | 3 month

SECONDARY OUTCOMES:
insulin sensitivity by a 3-hour hyperinsulinemic-euglycemic clamp, oral glucose tolerance test, liver fat and intramyocellular lipid by 1H-magnetic resonance spectroscopy. | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: SoJung Lee, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Yu WW, Lee S, Arslanian S, Tamim H, Kuk JL. Effects of Exercise on Resting Metabolic Rate in Adolescents with Overweight and Obesity. Child Obes. 2021 Jun;17(4):249-256. doi: 10.1089/chi.2020.0280. Epub 2021 Mar 18. PMID 33739874
- [Derived] Kuk JL, Lee S. Assessing the utility of cardiorespiratory fitness, visceral fat, and liver fat in predicting changes in insulin sensitivity beyond simple changes in body weight after exercise training in adolescents. Appl Physiol Nutr Metab. 2021 Jan;46(1):55-62. doi: 10.1139/apnm-2020-0284. Epub 2020 Jul 16. PMID 32674604
- [Derived] Kuk JL, Lee S. Sex and Ethnic Differences in the Relationship between Changes in Anthropometric Measurements and Visceral Fat in Adolescents with Obesity. J Pediatr. 2019 Oct;213:121-127. doi: 10.1016/j.jpeds.2019.05.052. Epub 2019 Jun 22. PMID 31235380